CLINICAL TRIAL: NCT03136484
Title: Efficacy and Safety of Semaglutide Versus Canagliflozin as add-on to Metformin in Subjects With Type 2 Diabetes
Acronym: SUSTAIN 8
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NN9535-4270; 2016-000989-35 (EudraCT Number); U1111-1180-3651 (Other: World Health Organization (WHO))
Record Dates: First submitted 2017-03-14; First posted 2017-05-02 (Actual); Results first posted 2019-12-17 (Actual); Last update posted 2020-01-21 (Actual); Status verified 2020-01

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — semaglutide; Canagliflozin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Semaglutide + canagliflozin placebo (Experimental)
  Interventions: Drug: Semaglutide; Drug: Placebo (canagliflozin)
- Canagliflozin + semaglutide placebo (Active Comparator)
  Interventions: Drug: Canagliflozin; Drug: Placebo (semaglutide)

INTERVENTIONS:
Drug: Semaglutide — Following a dose escalation phase of 8 weeks, semaglutide 1.0 mg once-weekly(administered subcutaneously, s.c., under the skin) and canagliflozin placebo once-daily (administered orally, as a tablet). Subjects will continue on their pre-trial daily dose of metformin.
  Arms: Semaglutide + canagliflozin placebo
Drug: Canagliflozin — Following a dose escalation phase of 8 weeks, canagliflozin 300 mg once-daily (administered orally, as a tablet) and semaglutide placebo (administered subcutaneously, s.c., under the skin). Subjects will continue on their pre-trial daily dose of metformin.
  Arms: Canagliflozin + semaglutide placebo
Drug: Placebo (canagliflozin) — Following a dose escalation phase of 8 weeks, semaglutide 1.0 mg once-weekly(administered subcutaneously, s.c., under the skin) and canagliflozin placebo once-daily (administered orally, as a tablet). Subjects will continue on their pre-trial daily dose of metformin.
  Arms: Semaglutide + canagliflozin placebo
Drug: Placebo (semaglutide) — Following a dose escalation phase of 8 weeks, canagliflozin 300 mg once-daily (administered orally, as a tablet) and semaglutide placebo (administered subcutaneously, s.c., under the skin). Subjects will continue on their pre-trial daily dose of metformin.
  Arms: Canagliflozin + semaglutide placebo

SUMMARY:
This trial is conducted in Africa, Asia, Europe, North and South America. The aim of the trial is to compare the effect of once-weekly (OW) dosing of subcutaneous semaglutide (1.0 mg) versus once-daily dosing of oral canagliflozin (300 mg) on glycaemic control in subjects with type 2 diabetes (T2D) on a background treatment of metformin

ELIGIBILITY:
Inclusion Criteria: - Informed consent obtained before any trial-related activities. Trial-related activities are any procedures that are carried out as part of the trial, including activities to determine suitability for the trial - Male or female, age equal to or above18 years at the time of signing informed consent - Diagnosed with type 2 diabetes mellitus (T2D) - HbA1c of 7.0-10.5% (53-91 mmol/mol, both inclusive) - Stable daily dose of metformin (equal to or above1500 mg or maximum tolerated dose as documented in the subject medical record and in compliance with current local label) for at least 90 days prior to the day of screening Exclusion Criteria: - Known or suspected hypersensitivity to trial product(s) or related products - Previous participation in this trial. Participation is defined as signed informed consent - Female who is pregnant, breast-feeding or intends to become pregnant or is of child-bearing potential and not using an adequate contraceptive method (adequate contraceptive measure as required by local regulation or practice) - Participation in any clinical trial of an approved or non-approved investigational medicinal product within 90 days prior to the day of screening - Any disorder which in the investigator's opinion might jeopardise subject's safety or compliance with the protocol - Subject with alanine aminotransferase (ALT) above 2.5 x upper normal limit (UNL) - Family or personal history of multiple endocrine neoplasia type 2 or medullary thyroid carcinoma. Family is defined as a first degree relative - History or presence of pancreatitis (acute or chronic) - History of diabetic ketoacidosis (DKA) - Any of the following: myocardial infarction (MI), stroke, hospitalization for unstable angina or transient ischaemic attack within the past 180 days prior to the day of screening - Subjects presently classified as being in New York Heart Association (NYHA) Class IV - Planned coronary, carotid or peripheral artery revascularisation known on the day of screening - Renal impairment measured as eGFR below 60 ml/min/1.73 m^2 as defined by Kidney Disease Improving global outcomes (KDIGO 2012) classification using isotope dilution mass spectrometry (IDMS) for serum creatinine measured at screening - Treatment with any medication for the indication of diabetes or obesity other than stated in the inclusion criteria within the past 90 days prior to the day of screening. However, short term insulin treatment for a maximum of 14 days prior to the day of screening is allowed - Proliferative retinopathy or maculopathy requiring acute treatment. Verified by fundus photography or dilated fundoscopy performed within the past 90 days prior to randomisation - Presence or history of malignant neoplasms within the past 5 years prior to the day of screening. Basal and squamous cell skin cancer and any carcinoma in-situ is allowed - Medical history of diabetes-related lower limb amputations or signs of critical lower limb ischemia, (e.g. skin ulcer, osteomyelitis, or gangrene) within the last 26 weeks prior to screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 788 (Actual)
Dates: Start 2017-03-15 (Actual); Primary Completion 2018-10-16 (Actual); Study Completion 2018-11-16 (Actual)

CONTACTS AND LOCATIONS:
Locations (102):
- United States (46):
  - Novo Nordisk Investigational Site, Anaheim, California
  - Novo Nordisk Investigational Site, La Mesa, California
  - Novo Nordisk Investigational Site, Los Angeles, California
  - Novo Nordisk Investigational Site, Montclair, California
  - Novo Nordisk Investigational Site, San Diego, California
  - Novo Nordisk Investigational Site, Spring Valley, California
  - Novo Nordisk Investigational Site, Tustin, California
  - Novo Nordisk Investigational Site, Walnut Creek, California
  - Novo Nordisk Investigational Site, Fleming Island, Florida
  - Novo Nordisk Investigational Site, Hallandale, Florida
  - Novo Nordisk Investigational Site, Hialeah, Florida
  - Novo Nordisk Investigational Site, Miami, Florida
  - Novo Nordisk Investigational Site, Spring Hill, Florida
  - Novo Nordisk Investigational Site, Conyers, Georgia
  - Novo Nordisk Investigational Site, Marietta, Georgia
  - Novo Nordisk Investigational Site, Meridian, Idaho
  - Novo Nordisk Investigational Site, Council Bluffs, Iowa
  - Novo Nordisk Investigational Site, Lexington, Kentucky
  - Novo Nordisk Investigational Site, Lake Charles, Louisiana
  - Novo Nordisk Investigational Site, Metairie, Louisiana
  - Novo Nordisk Investigational Site, Baltimore, Maryland
  - Novo Nordisk Investigational Site, Hyattsville, Maryland
  - Novo Nordisk Investigational Site, Detroit, Michigan
  - Novo Nordisk Investigational Site, Flint, Michigan
  - Novo Nordisk Investigational Site, Sterling Heights, Michigan
  - Novo Nordisk Investigational Site, Troy, Michigan
  - Novo Nordisk Investigational Site, Trenton, New Jersey
  - Novo Nordisk Investigational Site, Brooklyn, New York
  - Novo Nordisk Investigational Site, New Windsor, New York
  - Novo Nordisk Investigational Site, Greensboro, North Carolina
  - Novo Nordisk Investigational Site, Cincinnati, Ohio
  - Novo Nordisk Investigational Site, Maumee, Ohio
  - Novo Nordisk Investigational Site, Toledo, Ohio
  - Novo Nordisk Investigational Site, Corvallis, Oregon
  - Novo Nordisk Investigational Site, Anderson, South Carolina
  - Novo Nordisk Investigational Site, Amarillo, Texas
  - Novo Nordisk Investigational Site, Corpus Christi, Texas
  - Novo Nordisk Investigational Site, Dallas, Texas
  - Novo Nordisk Investigational Site, Houston, Texas
  - Novo Nordisk Investigational Site, Katy, Texas
  - Novo Nordisk Investigational Site, San Antonio, Texas
  - Novo Nordisk Investigational Site, Splendora, Texas
  - Novo Nordisk Investigational Site, St. George, Utah
  - Novo Nordisk Investigational Site, Herndon, Virginia
  - Novo Nordisk Investigational Site, Olympia, Washington
  - Novo Nordisk Investigational Site, Wenatchee, Washington
- Argentina (4):
  - Novo Nordisk Investigational Site, Buenos Aires
  - Novo Nordisk Investigational Site, CABA
  - Novo Nordisk Investigational Site, Rosario
  - Novo Nordisk Investigational Site, Salta
- Brazil (2):
  - Novo Nordisk Investigational Site, Porto Alegre
  - Novo Nordisk Investigational Site, Rio de Janeiro
- Canada (7):
  - Novo Nordisk Investigational Site, Surrey, British Columbia
  - Novo Nordisk Investigational Site, Brampton, Ontario
  - Novo Nordisk Investigational Site, Burlington, Ontario
  - Novo Nordisk Investigational Site, London, Ontario
  - Novo Nordisk Investigational Site, Sarnia, Ontario
  - Novo Nordisk Investigational Site, Toronto, Ontario
  - Novo Nordisk Investigational Site, Pointe-Claire, Quebec
- India (9):
  - Novo Nordisk Investigational Site, Hyderabad, Andhra Pradesh
  - Novo Nordisk Investigational Site, Rohtak, Haryana
  - Novo Nordisk Investigational Site, Bangalore, Karnataka
  - Novo Nordisk Investigational Site, Kochi, Kerala
  - Novo Nordisk Investigational Site, Mumbai, Maharashtra
  - Novo Nordisk Investigational Site, Nagpur, Maharashtra
  - Novo Nordisk Investigational Site, Jaipur, Rajasthan
  - Novo Nordisk Investigational Site, Chennai, Tamil Nadu
  - Novo Nordisk Investigational Site, Kolkata, West Bengal
- Ireland (3):
  - Novo Nordisk Investigational Site, Dublin
  - Novo Nordisk Investigational Site, Galway
  - Novo Nordisk Investigational Site, Mallow
- Novo Nordisk Investigational Site, Milan, Italy
- Lebanon (5):
  - Novo Nordisk Investigational Site, El Achrafiyé
  - Novo Nordisk Investigational Site, Hazmiyeh
  - Novo Nordisk Investigational Site, Lebanon - Beirut
  - Novo Nordisk Investigational Site, Mansourieh
  - Novo Nordisk Investigational Site, Zghartā
- Malaysia (6):
  - Novo Nordisk Investigational Site, Alor Gajah
  - Novo Nordisk Investigational Site, George Town
  - Novo Nordisk Investigational Site, Ipoh
  - Novo Nordisk Investigational Site, Malacca
  - Novo Nordisk Investigational Site, Sandakan
  - Novo Nordisk Investigational Site, Seremban
- Mexico (3):
  - Novo Nordisk Investigational Site, Cuernavaca, Morelos
  - Novo Nordisk Investigational Site, Mexico City, México, D.F.
  - Novo Nordisk Investigational Site, Monterrey, Nuevo León
- Sweden (5):
  - Novo Nordisk Investigational Site, Eksjö
  - Novo Nordisk Investigational Site, Kristianstad
  - Novo Nordisk Investigational Site, Lund
  - Novo Nordisk Investigational Site, Malmo
  - Novo Nordisk Investigational Site, Örebro
- United Kingdom (11):
  - Novo Nordisk Investigational Site, Basingstoke
  - Novo Nordisk Investigational Site, Bradford-on-Avon
  - Novo Nordisk Investigational Site, Dundee
  - Novo Nordisk Investigational Site, Haxey
  - Novo Nordisk Investigational Site, Nottingham
  - Novo Nordisk Investigational Site, Plymouth
  - Novo Nordisk Investigational Site, Soham
  - Novo Nordisk Investigational Site, Southampton
  - Novo Nordisk Investigational Site, Stevenage
  - Novo Nordisk Investigational Site, Torquay
  - Novo Nordisk Investigational Site, Wellingborough

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com

REFERENCES:
- [Result] Lingvay I, Catarig AM, Frias JP, Kumar H, Lausvig NL, le Roux CW, Thielke D, Viljoen A, McCrimmon RJ. Efficacy and safety of once-weekly semaglutide versus daily canagliflozin as add-on to metformin in patients with type 2 diabetes (SUSTAIN 8): a double-blind, phase 3b, randomised controlled trial. Lancet Diabetes Endocrinol. 2019 Nov;7(11):834-844. doi: 10.1016/S2213-8587(19)30311-0. Epub 2019 Sep 17. PMID 31540867
- [Result] McCrimmon RJ, Catarig AM, Frias JP, Lausvig NL, le Roux CW, Thielke D, Lingvay I. Effects of once-weekly semaglutide vs once-daily canagliflozin on body composition in type 2 diabetes: a substudy of the SUSTAIN 8 randomised controlled clinical trial. Diabetologia. 2020 Mar;63(3):473-485. doi: 10.1007/s00125-019-05065-8. Epub 2020 Jan 2. PMID 31897524
- [Derived] Natale P, Green SC, Tunnicliffe DJ, Pellegrino G, Toyama T, Strippoli GF. Glucagon-like peptide 1 (GLP-1) receptor agonists for people with chronic kidney disease and diabetes. Cochrane Database Syst Rev. 2025 Feb 18;2(2):CD015849. doi: 10.1002/14651858.CD015849.pub2. PMID 39963952
- [Derived] Pulleyblank R, Larsen NB. Cost-Effectiveness of Semaglutide vs. Empagliflozin, Canagliflozin, and Sitagliptin for Treatment of Patients with Type 2 Diabetes in Denmark: A Decision-Analytic Modelling Study. Pharmacoecon Open. 2023 Jul;7(4):579-591. doi: 10.1007/s41669-023-00416-z. Epub 2023 May 13. PMID 37178435
- [Derived] Lingvay I, Capehorn MS, Catarig AM, Johansen P, Lawson J, Sandberg A, Shaw R, Paine A. Efficacy of Once-Weekly Semaglutide vs Empagliflozin Added to Metformin in Type 2 Diabetes: Patient-Level Meta-analysis. J Clin Endocrinol Metab. 2020 Dec 1;105(12):e4593-604. doi: 10.1210/clinem/dgaa577. PMID 32827435

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was conducted at 115 sites in Argentina (5), Brazil (2), Canada (8), India (10), Ireland (4), Lebanon (5), Malaysia (5), Mexico (2), Sweden (5), United Kingdom (11) and United States (58).
Pre-assignment Details: Study design: Body composition (sub-study) was measured using dual x-ray absorptiometry (DXA) scans in a planned subset of randomised participants.
Groups:
- Semaglutide + Canagliflozin Placebo: Participants received subcutaneous (s.c.) injection of semaglutide once-weekly for 52 weeks: 0.25 milligrams (mg) during 0-4 weeks followed by 0.5 mg during 5-8 weeks and then 1.0 mg during 9-52 weeks. Participants also received placebo matched to canagliflozin tablet once-daily for 52 weeks.
- Canagliflozin + Semaglutide Placebo: Participants received canagliflozin tablet once-daily orally for 52 weeks: 100 mg tablet during 0-8 weeks followed by 300 mg tablet during 9-52 weeks. Participants also received placebo matched to semaglutide s.c. injection once-weekly for 52 weeks.
Period: Overall Study
Arm/Group | Semaglutide + Canagliflozin Placebo | Canagliflozin + Semaglutide Placebo
Started | 394 | 394
Exposed | 392 | 394
Completed | 367 | 372
Not Completed | 27 | 22
Not completed — Withdrawal by Subject | 19 | 14
Not completed — Lost to Follow-up | 7 | 8
Not completed — Death | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Semaglutide + Canagliflozin Placebo: Participants received s.c. injection of semaglutide once-weekly for 52 weeks: 0.25 milligrams (mg) during 0-4 weeks followed by 0.5 mg during 5-8 weeks and then 1.0 mg during 9-52 weeks. Participants also received placebo matched to canagliflozin tablet once-daily for 52 weeks.
- Total: Total of all reporting groups
Arm/Group | Semaglutide + Canagliflozin Placebo | Canagliflozin + Semaglutide Placebo | Total
Number analyzed (Participants) | 394 | 394 | 788
Age, Continuous [Mean (Standard Deviation); unit: Years] | 55.7 (11.1) | 57.5 (10.7) | 56.6 (10.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 171 | 193 | 364
  Male | 223 | 201 | 424
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 156 | 137 | 293
  Not Hispanic or Latino | 238 | 257 | 495
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: Participants]
  Race : American Indian or Alaska native | 1 | 3 | 4
  Race : Asian | 62 | 63 | 125
  Race : Black or African American | 28 | 30 | 58
  Race : Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Race : White | 297 | 290 | 587
  Race : Other | 6 | 7 | 13
  Race : Not Applicable | 0 | 1 | 1
HbA1c [Mean (Standard Deviation); unit: Percentage (%) of HbA1c] | 8.3 (1.0) | 8.2 (1.0) | 8.3 (1.0)

OUTCOME MEASURES:

1. Primary Outcome: Change in HbA1c
Description: Change from baseline (week 0) to week 52 in HbA1c (glycosylated haemoglobin) was evaluated. Results are based on the 'on-treatment without rescue medication' observation period, which started at the date of first dose to either the day of last dose plus 7 days or first initiation of rescue medication, whichever came first; and 'In-trial' observation period which started at the date of randomisation and include the period after initiation of rescue medication and/or premature trial product discontinuation, if any and ended at the last contact, withdrawal of consent or death, whichever came first.
Time Frame: Week 0, week 52
Population: Full analysis set comprised of all randomised participants. "Number analyzed"=participants with available data.
Measure: Mean (Standard Deviation); unit: Percentage (%) of HbA1c
Arm/Group | Semaglutide + Canagliflozin Placebo | Canagliflozin + Semaglutide Placebo
Number analyzed (Participants) | 394 | 394
Percentage (%) of HbA1c
  On-treatment without rescue medication: number analyzed (Participants) | 293 | 313
  On-treatment without rescue medication | -1.7 (1.1) | -1.0 (1.0)
  In-trial: number analyzed (Participants) | 361 | 362
  In-trial | -1.5 (1.3) | -1.0 (1.1)
Statistical Analysis 1: Comparison: Semaglutide + Canagliflozin Placebo vs Canagliflozin + Semaglutide Placebo; The responses were analysed using an analysis of covariance (ANCOVA) with treatment, region and stratification factor as fixed factors and baseline value as covariate. Before analysis, missing data were multiple imputed using observed data from participants within the same group defined by randomised treatment, using a regression model including region and stratification factor as categorical effects and data from baseline and all previous visits as covariates; Test type: Non-Inferiority — The non-inferiority p-value was calculated as two times the one-sided p-value from a t-distributed test statistic comparing the treatment contrast with 0.3 rather than zero as in a superiority test; p < .0001, ANCOVA; Treatment difference = -0.49, 95% CI 2-sided [-0.65 to -0.33] — Semaglutide + canagliflozin placebo vs Canagliflozin + semaglutide placebo
Statistical Analysis 2: Comparison: Semaglutide + Canagliflozin Placebo vs Canagliflozin + Semaglutide Placebo; The responses were analysed using an ANCOVA with treatment, region and stratification factor as fixed factors and baseline value as covariate. Before analysis, missing data were multiple imputed using observed data from participants within the same group defined by randomised treatment, using a regression model including region and stratification factor as categorical effects and data from baseline and all previous visits as covariates; Test type: Superiority; p < .0001, ANCOVA; Treatment difference = -0.49, 95% CI 2-sided [-0.65 to -0.33] — Semaglutide + canagliflozin placebo vs Canagliflozin + semaglutide placebo

2. Secondary Outcome: Change in Body Weight (kg)
Description: Change from baseline (week 0) to week 52 in body weight was evaluated. Results are based on the 'on-treatment without rescue medication' observation period, which started at the date of first dose to either the day of last dose plus 7 days or first initiation of rescue medication, whichever came first.
Time Frame: Week 0, week 52
Population: Full analysis set comprised of all randomised participants. "Number analyzed"=participants with available data.
Measure: Mean (Standard Deviation); unit: Kilogram (kg)
Arm/Group | Semaglutide + Canagliflozin Placebo | Canagliflozin + Semaglutide Placebo
Number analyzed (Participants) | 394 | 394
Kilogram (kg) | -5.7 (5.4) | -4.3 (4.0)

3. Secondary Outcome: Change in Total Fat Mass (kg)
Description: Change from baseline (week 0) to week 52 in total fat mass was evaluated. Results are based on the 'on-treatment without rescue medication' observation period, which started at the date of first dose to either the day of last dose plus 7 days or first initiation of rescue medication, whichever came first.
Time Frame: Week 0, week 52
Population: Dual X-ray absorptiometry (DXA) analysis set comprised of all randomised participants who are included in the body composition sub-study. "Number analyzed"=participants with available data.
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Semaglutide + Canagliflozin Placebo | Canagliflozin + Semaglutide Placebo
Number analyzed (Participants) | 88 | 90
kg | -3.72 (4.50) | -2.63 (3.30)

4. Secondary Outcome: Change in FPG (Fasting Plasma Glucose)
Description: Change from baseline (week 0) to week 52 in FPG was evaluated. Results are based on the 'on-treatment without rescue medication' observation period, which started at the date of first dose to either the day of last dose plus 7 days or first initiation of rescue medication, whichever came first.
Time Frame: Week 0, week 52
Population: Full analysis set comprised of all randomised participants. "Number analyzed"=participants with available data.
Measure: Mean (Standard Deviation); unit: Millimoles per liter (mmol/L)
Arm/Group | Semaglutide + Canagliflozin Placebo | Canagliflozin + Semaglutide Placebo
Number analyzed (Participants) | 394 | 394
Millimoles per liter (mmol/L) | -2.54 (2.77) | -2.00 (2.53)

5. Secondary Outcome: Change in SMPG (Self-measured Plasma Glucose)- Mean 7-point Profile
Description: Change from baseline (week 0) to week 52 in SMPG- mean 7-point profile was evaluated. SMPG was recorded at the following 7 time points: before breakfast, 90 minutes after start of breakfast, before lunch, 90 minutes after start of lunch, before dinner, 90 minutes after dinner and at bedtime. Mean 7-point profile was defined as the area under the profile, calculated using the trapezoidal method, divided by the measurement time. Results are based on the 'on-treatment without rescue medication' observation period, which started at the date of first dose to either the day of last dose plus 7 days or first initiation of rescue medication, whichever came first.
Time Frame: Week 0, week 52
Population: Full analysis set comprised of all randomised participants. "Number analyzed"=participants with available data.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Semaglutide + Canagliflozin Placebo | Canagliflozin + Semaglutide Placebo
Number analyzed (Participants) | 394 | 394
mmol/L | -2.8 (2.3) | -1.9 (2.7)

6. Secondary Outcome: Change in SMPG- Mean Postprandial Increment Over All Meals
Description: Change from baseline (week 0) to week 52 in SMPG- mean postprandial increment over all meals was evaluated. Results are based on the 'on-treatment without rescue medication' observation period, which started at the date of first dose to either the day of last dose plus 7 days or first initiation of rescue medication, whichever came first.
Time Frame: Week 0, week 52
Population: Full analysis set comprised of all randomised participants. "Number analyzed"=participants with available data.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Semaglutide + Canagliflozin Placebo | Canagliflozin + Semaglutide Placebo
Number analyzed (Participants) | 394 | 394
mmol/L | -0.6 (2.1) | -0.6 (2.0)

7. Secondary Outcome: Change in Fasting Total Cholesterol
Description: Change from baseline (week 0) to week 52 in fasting total cholesterol (mmol/L) is presented as ratio to baseline. Results are based on the 'on-treatment without rescue medication' observation period, which started at the date of first dose to either the day of last dose plus 7 days or first initiation of rescue medication, whichever came first.
Time Frame: Week 0, week 52
Population: Full analysis set comprised of all randomised participants. "Number analyzed"=participants with available data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of total cholesterol
Arm/Group | Semaglutide + Canagliflozin Placebo | Canagliflozin + Semaglutide Placebo
Number analyzed (Participants) | 394 | 394
Ratio of total cholesterol | 0.96 (19.3) | 1.03 (18.2)

8. Secondary Outcome: Change in Fasting LDL-cholesterol
Description: Change from baseline (week 0) to week 52 in fasting low-density lipoprotein (LDL) cholesterol (mmol/L) is presented as ratio to baseline. Results are based on the 'on-treatment without rescue medication' observation period, which started at the date of first dose to either the day of last dose plus 7 days or first initiation of rescue medication, whichever came first.
Time Frame: Week 0, week 52
Population: Full analysis set comprised of all randomised participants. "Number analyzed"=participants with available data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of LDL-cholesterol
Arm/Group | Semaglutide + Canagliflozin Placebo | Canagliflozin + Semaglutide Placebo
Number analyzed (Participants) | 394 | 394
Ratio of LDL-cholesterol | 0.96 (32.2) | 1.05 (29.0)

9. Secondary Outcome: Change in Fasting HDL-cholesterol
Description: Change from baseline (week 0) to week 52 in fasting high-density lipoprotein (HDL) cholesterol (mmol/L) is presented as ratio to baseline. Results are based on the 'on-treatment without rescue medication' observation period, which started at the date of first dose to either the day of last dose plus 7 days or first initiation of rescue medication, whichever came first.
Time Frame: Week 0, week 52
Population: Full analysis set comprised of all randomised participants. "Number analyzed"=participants with available data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of HDL-cholesterol
Arm/Group | Semaglutide + Canagliflozin Placebo | Canagliflozin + Semaglutide Placebo
Number analyzed (Participants) | 394 | 394
Ratio of HDL-cholesterol | 1.04 (13.1) | 1.08 (13.6)

10. Secondary Outcome: Change in Fasting Triglycerides
Description: Change from baseline (week 0) to week 52 in fasting triglycerides (mmol/L) is presented as ratio to baseline. Results are based on the 'on-treatment without rescue medication' observation period, which started at the date of first dose to either the day of last dose plus 7 days or first initiation of rescue medication, whichever came first.
Time Frame: Week 0, week 52
Population: Full analysis set comprised of all randomised participants. "Number analyzed"=participants with available data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of triglycerides
Arm/Group | Semaglutide + Canagliflozin Placebo | Canagliflozin + Semaglutide Placebo
Number analyzed (Participants) | 394 | 394
Ratio of triglycerides | 0.86 (40.6) | 0.92 (38.2)

11. Secondary Outcome: Change in Vital Signs (Systolic Blood Pressure and Diastolic Blood Pressure)
Description: Change from baseline (week 0) to week 52 in systolic blood pressure and diastolic blood pressure. Results are based on the 'on-treatment without rescue medication' observation period, which started at the date of first dose to either the day of last dose plus 7 days or first initiation of rescue medication, whichever came first.
Time Frame: Week 0, week 52
Population: Full analysis set comprised of all randomised participants. "Number analyzed"=participants with available data.
Measure: Mean (Standard Deviation); unit: Millimeters of mercury (mmHg)
Arm/Group | Semaglutide + Canagliflozin Placebo | Canagliflozin + Semaglutide Placebo
Number analyzed (Participants) | 394 | 394
Millimeters of mercury (mmHg)
  Systolic blood pressure: number analyzed (Participants) | 298 | 313
  Systolic blood pressure | -3.7 (14.0) | -5.8 (13.5)
  Diastolic blood pressure: number analyzed (Participants) | 298 | 313
  Diastolic blood pressure | -1.2 (9.8) | -2.9 (9.0)

12. Secondary Outcome: Percentage Change in Body Weight (%)
Description: as for outcome 2
Time Frame: Week 0, week 52
Population: Full analysis set comprised of all randomised participants. "Number analyzed"=participants with available data.
Measure: Mean (Standard Deviation); unit: Percentage change
Arm/Group | Semaglutide + Canagliflozin Placebo | Canagliflozin + Semaglutide Placebo
Number analyzed (Participants) | 394 | 394
Percentage change | -6.2 (6.1) | -4.7 (4.0)

13. Secondary Outcome: Change in Body Mass Index (BMI)
Description: Change from baseline (week 0) to week 52 in BMI was evaluated. Results are based on the 'on-treatment without rescue medication' observation period, which started at the date of first dose to either the day of last dose plus 7 days or first initiation of rescue medication, whichever came first.
Time Frame: Week 0, week 52
Population: Full analysis set comprised of all randomised participants. "Number analyzed"=participants with available data.
Measure: Mean (Standard Deviation); unit: Kilogram per square meter (kg/m^2)
Arm/Group | Semaglutide + Canagliflozin Placebo | Canagliflozin + Semaglutide Placebo
Number analyzed (Participants) | 394 | 394
Kilogram per square meter (kg/m^2) | -2.0 (2.0) | -1.5 (1.4)

14. Secondary Outcome: Change in Waist Circumference
Description: Change from baseline (week 0) to week 52 in waist circumference was evaluated. Results are based on the 'on-treatment without rescue medication' observation period, which started at the date of first dose to either the day of last dose plus 7 days or first initiation of rescue medication, whichever came first.
Time Frame: Week 0, week 52
Population: Full analysis set comprised of all randomised participants. "Number analyzed"=participants with available data.
Measure: Mean (Standard Deviation); unit: Centimeter (cm)
Arm/Group | Semaglutide + Canagliflozin Placebo | Canagliflozin + Semaglutide Placebo
Number analyzed (Participants) | 394 | 394
Centimeter (cm) | -4.2 (6.2) | -3.0 (5.4)

15. Secondary Outcome: Percentage Change in Total Fat Mass (%)
Description: as for outcome 3
Time Frame: Week 0, week 52
Population: DXA analysis set comprised of all randomised participants who are included in the body composition sub-study. "Number analyzed"=participants with available data.
Measure: Mean (Standard Deviation); unit: Percentage change
Arm/Group | Semaglutide + Canagliflozin Placebo | Canagliflozin + Semaglutide Placebo
Number analyzed (Participants) | 88 | 90
Percentage change | -1.55 (2.76) | -1.21 (2.64)

16. Secondary Outcome: Change in Total Lean Mass (kg)
Description: Change from baseline (week 0) to week 52 in total lean mass was evaluated. Results are based on the 'on-treatment without rescue medication' observation period, which started at the date of first dose to either the day of last dose plus 7 days or first initiation of rescue medication, whichever came first.
Time Frame: Week 0, week 52
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Semaglutide + Canagliflozin Placebo | Canagliflozin + Semaglutide Placebo
Number analyzed (Participants) | 88 | 90
kg | -2.06 (2.15) | -1.53 (2.21)

17. Secondary Outcome: Percentage Change in Total Lean Mass (%)
Description: as for outcome 16
Time Frame: Week 0, week 52
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: Percentage change
Arm/Group | Semaglutide + Canagliflozin Placebo | Canagliflozin + Semaglutide Placebo
Number analyzed (Participants) | 88 | 90
Percentage change | 1.38 (2.66) | 1.09 (2.56)

18. Secondary Outcome: Change in Visceral Fat Mass (kg)
Description: Change from baseline (week 0) to week 52 in visceral fat mass was evaluated. Results are based on the 'on-treatment without rescue medication' observation period, which started at the date of first dose to either the day of last dose plus 7 days or first initiation of rescue medication, whichever came first.
Time Frame: Week 0, week 52
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Semaglutide + Canagliflozin Placebo | Canagliflozin + Semaglutide Placebo
Number analyzed (Participants) | 88 | 90
kg | -0.20 (0.40) | -0.13 (0.32)

19. Secondary Outcome: Percentage Change in Visceral Fat Mass (%)
Description: as for outcome 18
Time Frame: Week 0, week 52
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: Percentage change
Arm/Group | Semaglutide + Canagliflozin Placebo | Canagliflozin + Semaglutide Placebo
Number analyzed (Participants) | 88 | 90
Percentage change | -0.81 (7.30) | 0.16 (4.36)

20. Secondary Outcome: Change in Ratio Between Total Fat Mass and Total Lean Mass
Description: Change from baseline (week 0) to week 52 in ratio between total fat mass and total lean mass was evaluated. Results are based on the 'on-treatment without rescue medication' observation period, which started at the date of first dose to either the day of last dose plus 7 days or first initiation of rescue medication, whichever came first.
Time Frame: Week 0, week 52
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: total fat mass/total lean mass ratio
Arm/Group | Semaglutide + Canagliflozin Placebo | Canagliflozin + Semaglutide Placebo
Number analyzed (Participants) | 88 | 90
total fat mass/total lean mass ratio | -0.04 (0.08) | -0.03 (0.07)

21. Secondary Outcome: Participants Who Achieved HbA1c < 7.0% (53 mmol/Mol), American Diabetes Association (ADA) Target (Yes/no)
Description: Percentage of participants who achieved HbA1c < 7.0% (53 millimoles per mole [mmol/mol]), ADA target (yes/no) is presented. Results are based on the 'on-treatment without rescue medication' observation period, which started at the date of first dose to either the day of last dose plus 7 days or first initiation of rescue medication, whichever came first.
Time Frame: Week 52
Population: Full analysis set comprised of all randomised participants. "Number analyzed"=participants with available data.
Measure: Number; unit: Percentage of participants
Arm/Group | Semaglutide + Canagliflozin Placebo | Canagliflozin + Semaglutide Placebo
Number analyzed (Participants) | 293 | 313
Percentage of participants
  Yes | 76.1 | 50.8
  No | 23.9 | 49.2

22. Secondary Outcome: Participants Who Achieved HbA1c ≤ 6.5% (48 mmol/Mol), American Association of Clinical Endocrinologists (AACE) Target (Yes/no)
Description: Percentage of participants who achieved HbA1c ≤ 6.5% (48 mmol/mol), AACE target (yes/no) is presented. Results are based on the 'on-treatment without rescue medication' observation period, which started at the date of first dose to either the day of last dose plus 7 days or first initiation of rescue medication, whichever came first.
Time Frame: Week 52
Population: Full analysis set comprised of all randomised participants. "Number analyzed"=participants with available data.
Measure: Number; unit: Percentage of participants
Arm/Group | Semaglutide + Canagliflozin Placebo | Canagliflozin + Semaglutide Placebo
Number analyzed (Participants) | 293 | 313
Percentage of participants
  Yes | 62.1 | 26.8
  No | 37.9 | 73.2

23. Secondary Outcome: Participants Who Achieved HbA1c Reduction ≥1% (Yes/no)
Description: Percentage of participants who achieved ≥1% reduction of baseline HbA1c (yes/no) is presented. Results are based on the 'on-treatment without rescue medication' observation period, which started at the date of first dose to either the day of last dose plus 7 days or first initiation of rescue medication, whichever came first.
Time Frame: Week 0, week 52
Population: Full analysis set comprised of all randomised participants. "Number analyzed"=participants with available data.
Measure: Number; unit: Percentage of participants
Arm/Group | Semaglutide + Canagliflozin Placebo | Canagliflozin + Semaglutide Placebo
Number analyzed (Participants) | 293 | 313
Percentage of participants
  Yes | 76.5 | 48.6
  No | 23.5 | 51.4

24. Secondary Outcome: Participants Who Achieved Weight Loss ≥3% (Yes/no)
Description: Percentage of participants losing ≥3% of baseline body weight (yes/no) is presented. Results are based on the 'on-treatment without rescue medication' observation period, which started at the date of first dose to either the day of last dose plus 7 days or first initiation of rescue medication, whichever came first.
Time Frame: Week 0, week 52
Population: Full analysis set comprised of all randomised participants. "Number analyzed"=participants with available data.
Measure: Number; unit: Percentage of participants
Arm/Group | Semaglutide + Canagliflozin Placebo | Canagliflozin + Semaglutide Placebo
Number analyzed (Participants) | 298 | 313
Percentage of participants
  Yes | 68.8 | 64.9
  No | 31.2 | 35.1

25. Secondary Outcome: Participants Who Achieved Weight Loss ≥5% (Yes/no)
Description: Percentage of participants losing ≥5% of baseline body weight (yes/no) is presented. Results are based on the 'on-treatment without rescue medication' observation period, which started at the date of first dose to either the day of last dose plus 7 days or first initiation of rescue medication, whichever came first.
Time Frame: Week 0, week 52
Population: Full analysis set comprised of all randomised participants. "Number analyzed"=participants with available data.
Measure: Number; unit: Percentage of participants
Arm/Group | Semaglutide + Canagliflozin Placebo | Canagliflozin + Semaglutide Placebo
Number analyzed (Participants) | 298 | 313
Percentage of participants
  Yes | 52.7 | 47.0
  No | 47.3 | 53.0

26. Secondary Outcome: Participants Who Achieved Weight Loss ≥10% (Yes/no)
Description: Percentage of participants losing ≥10% of baseline body weight is presented. Results are based on the 'on-treatment without rescue medication' observation period, which started at the date of first dose to either the day of last dose plus 7 days or first initiation of rescue medication, whichever came first.
Time Frame: Week 0, week 52
Population: Full analysis set comprised of all randomised participants. "Number analyzed"=participants with available data.
Measure: Number; unit: Percentage of participants
Arm/Group | Semaglutide + Canagliflozin Placebo | Canagliflozin + Semaglutide Placebo
Number analyzed (Participants) | 298 | 313
Percentage of participants
  Yes | 23.2 | 8.9
  No | 76.8 | 91.1

27. Secondary Outcome: Participants Who Achieved HbA1c Below 7.0% (53 mmol/Mol) Without Severe or Blood Glucose (BG)-Confirmed Symptomatic Hypoglycaemia Episodes and no Weight Gain (Yes/no)
Description: Severe or BG-confirmed symptomatic hypoglycaemia is an episode that is severe according to the American Diabetes Association classification or blood glucose-confirmed by a plasma glucose value <3.1 mmol/L (56 milligrams per deciliter [mg/dL]) with symptoms consistent with hypoglycaemia. Percentage of participants who achieved HbA1c below 7.0% (53 mmol/mol) without severe or blood glucose confirmed symptomatic hypoglycaemia episodes and no weight gain (yes/no) is presented. Results are based on the 'on-treatment without rescue medication' observation period, which started at the date of first dose to either the day of last dose plus 7 days or first initiation of rescue medication, whichever came first.
Time Frame: Week 0, week 52
Population: Full analysis set comprised of all randomised participants. "Number analyzed"=participants with available data.
Measure: Number; unit: Percentage of participants
Arm/Group | Semaglutide + Canagliflozin Placebo | Canagliflozin + Semaglutide Placebo
Number analyzed (Participants) | 293 | 313
Percentage of participants
  Yes | 69.6 | 45.0
  No | 30.4 | 55.0

28. Secondary Outcome: Participants Who Achieved HbA1c Reduction ≥1% and Weight Loss ≥3% (Yes/no)
Description: Percentage of participants who achieved ≥1% reduction of baseline HbA1c and losing ≥3% of baseline body weight (yes/no) is presented. Results are based on the 'on-treatment without rescue medication' observation period, which started at the date of first dose to either the day of last dose plus 7 days or first initiation of rescue medication, whichever came first.
Time Frame: Week 0, week 52
Population: Full analysis set comprised of all randomised participants. "Number analyzed"=participants with available data.
Measure: Number; unit: Percentage of participants
Arm/Group | Semaglutide + Canagliflozin Placebo | Canagliflozin + Semaglutide Placebo
Number analyzed (Participants) | 293 | 313
Percentage of participants
  Yes | 57.3 | 34.8
  No | 42.7 | 65.2

29. Secondary Outcome: Participants Who Achieved HbA1c Reduction ≥1% and Weight Loss ≥5% (Yes/no)
Description: Percentage of participants who achieved ≥1% reduction of baseline HbA1c and losing ≥5% of baseline body weight (yes/no) is presented. Results are based on the 'on-treatment without rescue medication' observation period, which started at the date of first dose to either the day of last dose plus 7 days or first initiation of rescue medication, whichever came first.
Time Frame: Week 0, week 52
Population: Full analysis set comprised of all randomised participants. "Number analyzed"=participants with available data.
Measure: Number; unit: Percentage of participants
Arm/Group | Semaglutide + Canagliflozin Placebo | Canagliflozin + Semaglutide Placebo
Number analyzed (Participants) | 293 | 313
Percentage of participants
  Yes | 45.1 | 25.9
  No | 54.9 | 74.1

30. Secondary Outcome: Participants Who Achieved HbA1c Reduction ≥1% and Weight Loss ≥10% (Yes/no)
Description: Percentage of participants who achieved ≥1% reduction of baseline HbA1c and losing ≥10% of baseline body weight (yes/no) is presented. Results are based on the 'on-treatment without rescue medication' observation period, which started at the date of first dose to either the day of last dose plus 7 days or first initiation of rescue medication, whichever came first.
Time Frame: Week 0, week 52
Population: Full analysis set comprised of all randomised participants. "Number analyzed"=participants with available data.
Measure: Number; unit: Percentage of participants
Arm/Group | Semaglutide + Canagliflozin Placebo | Canagliflozin + Semaglutide Placebo
Number analyzed (Participants) | 293 | 313
Percentage of participants
  Yes | 21.8 | 6.1
  No | 78.2 | 93.9

31. Secondary Outcome: Total Number of Treatment Emergent Adverse Events (TEAEs)
Description: A TEAE is defined as an adverse event with onset in the on-treatment observation period (which started at the date of first dose of trial product and included the period after initiation of rescue medication, if any and excluded the period after premature trial product discontinuation, if any. TEAEs assessed up to approximately 57 weeks is presented.
Time Frame: Weeks 0-57
Population: Safety analysis set comprised of participants exposed to at least one dose of trial product.
Measure: Number; unit: Adverse events
Arm/Group | Semaglutide + Canagliflozin Placebo | Canagliflozin + Semaglutide Placebo
Number analyzed (Participants) | 392 | 394
Adverse events | 1189 | 1138

32. Secondary Outcome: Change in Haematological Parameter- Haemoglobin
Description: Change from baseline (week 0) to week 52 in haemoglobin (mmol/L) is presented as ratio to baseline. Results are based on the 'on-treatment' observation period which started at the date of first dose of trial product and include the period after initiation of rescue medication, if any and excludes the period after premature trial product discontinuation, if any.
Time Frame: Week 0, week 52
Population: Safety analysis set comprised of participants exposed to at least one dose of trial product. "Number analyzed"=participants with available data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of haemoglobin
Arm/Group | Semaglutide + Canagliflozin Placebo | Canagliflozin + Semaglutide Placebo
Number analyzed (Participants) | 392 | 394
Ratio of haemoglobin | 0.99 (8.0) | 1.05 (8.5)

33. Secondary Outcome: Change in Haematological Parameter- Haematocrit
Description: Change from baseline (week 0) to week 52 in haematocrit (%) is presented as ratio to baseline. Results are based on the 'on-treatment' observation period which started at the date of first dose of trial product and include the period after initiation of rescue medication, if any and excludes the period after premature trial product discontinuation, if any.
Time Frame: Week 0, week 52
Population: as for outcome 32
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of haematocrit
Arm/Group | Semaglutide + Canagliflozin Placebo | Canagliflozin + Semaglutide Placebo
Number analyzed (Participants) | 392 | 394
Ratio of haematocrit | 0.99 (6.8) | 1.04 (6.9)

34. Secondary Outcome: Change in Haematological Parameter- Erythrocytes
Description: Change from baseline (week 0) to week 52 in erythrocytes (10^12 cells/L) is presented as ratio to baseline. Results are based on the 'on-treatment' observation period which started at the date of first dose of trial product and include the period after initiation of rescue medication, if any and excludes the period after premature trial product discontinuation, if any.
Time Frame: Week 0, week 52
Population: as for outcome 32
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of erythrocytes
Arm/Group | Semaglutide + Canagliflozin Placebo | Canagliflozin + Semaglutide Placebo
Number analyzed (Participants) | 392 | 394
Ratio of erythrocytes | 0.99 (5.7) | 1.04 (6.0)

35. Secondary Outcome: Change in Haematological Parameter- Leukocytes
Description: Change from baseline (week 0) to week 52 in leukocytes (10^9 cells/L) is presented as ratio to baseline. Results are based on the 'on-treatment' observation period which started at the date of first dose of trial product and include the period after initiation of rescue medication, if any and excludes the period after premature trial product discontinuation, if any.
Time Frame: Week 0, week 52
Population: as for outcome 32
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of leukocytes
Arm/Group | Semaglutide + Canagliflozin Placebo | Canagliflozin + Semaglutide Placebo
Number analyzed (Participants) | 392 | 394
Ratio of leukocytes | 0.97 (20.3) | 0.98 (17.5)

36. Secondary Outcome: Change in Haematological Parameter- Thrombocytes
Description: Change from baseline (week 0) to week 52 in thrombocytes (10^9 cells/L) is presented as ratio to baseline. Results are based on the 'on-treatment' observation period which started at the date of first dose of trial product and include the period after initiation of rescue medication, if any and excludes the period after premature trial product discontinuation, if any.
Time Frame: Week 0, week 52
Population: as for outcome 32
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of thrombocytes
Arm/Group | Semaglutide + Canagliflozin Placebo | Canagliflozin + Semaglutide Placebo
Number analyzed (Participants) | 392 | 394
Ratio of thrombocytes | 1.04 (14.4) | 1.00 (15.4)

37. Secondary Outcome: Change in Biochemistry Parameter- Amylase
Description: Change from baseline (week 0) to week 52 in amylase (units per liter [U/L]) is presented as ratio to baseline. Results are based on the 'on-treatment' observation period which started at the date of first dose of trial product and include the period after initiation of rescue medication, if any and excludes the period after premature trial product discontinuation, if any.
Time Frame: Week 0, week 52
Population: as for outcome 32
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of amylase
Arm/Group | Semaglutide + Canagliflozin Placebo | Canagliflozin + Semaglutide Placebo
Number analyzed (Participants) | 392 | 394
Ratio of amylase | 1.16 (26.5) | 1.09 (24.4)

38. Secondary Outcome: Change in Biochemistry Parameter- Lipase
Description: Change from baseline (week 0) to week 52 in lipase (U/L) is presented as ratio to baseline. Results are based on the 'on-treatment' observation period which started at the date of first dose of trial product and include the period after initiation of rescue medication, if any and excludes the period after premature trial product discontinuation, if any.
Time Frame: Week 0, week 52
Population: as for outcome 32
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of lipase
Arm/Group | Semaglutide + Canagliflozin Placebo | Canagliflozin + Semaglutide Placebo
Number analyzed (Participants) | 392 | 394
Ratio of lipase | 1.25 (54.5) | 1.01 (51.5)

39. Secondary Outcome: Change in Biochemistry Parameter- ALT
Description: Change from baseline (week 0) to week 52 in alanine aminotransferase (ALT) (U/L) is presented as ratio to baseline. Results are based on the 'on-treatment' observation period which started at the date of first dose of trial product and include the period after initiation of rescue medication, if any and excludes the period after premature trial product discontinuation, if any.
Time Frame: Week 0, week 52
Population: as for outcome 32
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of ALT
Arm/Group | Semaglutide + Canagliflozin Placebo | Canagliflozin + Semaglutide Placebo
Number analyzed (Participants) | 392 | 394
Ratio of ALT | 0.79 (49.5) | 0.79 (45.3)

40. Secondary Outcome: Change in Biochemistry Parameter- AST
Description: Change from baseline (week 0) to week 52 in aspartate aminotransferase (AST) (U/L) is presented as ratio to baseline. Results are based on the 'on-treatment' observation period which started at the date of first dose of trial product and include the period after initiation of rescue medication, if any and excludes the period after premature trial product discontinuation, if any.
Time Frame: Week 0, week 52
Population: as for outcome 32
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of AST
Arm/Group | Semaglutide + Canagliflozin Placebo | Canagliflozin + Semaglutide Placebo
Number analyzed (Participants) | 392 | 394
Ratio of AST | 0.89 (37.5) | 0.86 (37.4)

41. Secondary Outcome: Change in Biochemistry Parameter- ALP
Description: Change from baseline (week 0) to week 52 in alkaline phosphatase (ALP) (U/L) is presented as ratio to baseline. Results are based on the 'on-treatment' observation period which started at the date of first dose of trial product and include the period after initiation of rescue medication, if any and excludes the period after premature trial product discontinuation, if any.
Time Frame: Week 0, week 52
Population: as for outcome 32
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of ALP
Arm/Group | Semaglutide + Canagliflozin Placebo | Canagliflozin + Semaglutide Placebo
Number analyzed (Participants) | 392 | 394
Ratio of ALP | 0.96 (19.6) | 0.95 (16.8)

42. Secondary Outcome: Change in Biochemistry Parameter- Total Bilirubin
Description: Change from baseline (week 0) to week 52 in total bilirubin (U/L) is presented as ratio to baseline. Results are based on the 'on-treatment' observation period which started at the date of first dose of trial product and include the period after initiation of rescue medication, if any and excludes the period after premature trial product discontinuation, if any.
Time Frame: Week 0, week 52
Population: as for outcome 32
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of total bilirubin
Arm/Group | Semaglutide + Canagliflozin Placebo | Canagliflozin + Semaglutide Placebo
Number analyzed (Participants) | 392 | 394
Ratio of total bilirubin | 1.06 (32.1) | 1.13 (33.9)

43. Secondary Outcome: Change in Biochemistry Parameter- Creatinine
Description: Change from baseline (week 0) to week 52 in creatinine (micromoles per liter [umol/L]) is presented as ratio to baseline. Results are based on the 'on-treatment' observation period which started at the date of first dose of trial product and include the period after initiation of rescue medication, if any and excludes the period after premature trial product discontinuation, if any.
Time Frame: Week 0, week 52
Population: as for outcome 32
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of creatinine
Arm/Group | Semaglutide + Canagliflozin Placebo | Canagliflozin + Semaglutide Placebo
Number analyzed (Participants) | 392 | 394
Ratio of creatinine | 1.03 (11.0) | 1.04 (11.9)

44. Secondary Outcome: Change in Biochemistry Parameter- eGFR
Description: Estimated glomerular filtration rate (eGFR) (milliliters per minute per 1.73 square meters [mL/min/1.73m^2])is calculated using the equation from the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI). Change from baseline (week 0) to week 52 in eGFR is presented as ratio to baseline. Results are based on the 'on-treatment' observation period which started at the date of first dose of trial product and include the period after initiation of rescue medication, if any and excludes the period after premature trial product discontinuation, if any.
Time Frame: Week 0, week 52
Population: as for outcome 32
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of eGFR
Arm/Group | Semaglutide + Canagliflozin Placebo | Canagliflozin + Semaglutide Placebo
Number analyzed (Participants) | 392 | 394
Ratio of eGFR | 0.98 (8.4) | 0.96 (9.7)

45. Secondary Outcome: Change in Biochemistry Parameter- Albumin
Description: Change from baseline (week 0) to week 52 in albumin (g/dL) is presented as ratio to baseline. Results are based on the 'on-treatment' observation period which started at the date of first dose of trial product and include the period after initiation of rescue medication, if any and excludes the period after premature trial product discontinuation, if any.
Time Frame: Week 0, week 52
Population: as for outcome 32
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of albumin
Arm/Group | Semaglutide + Canagliflozin Placebo | Canagliflozin + Semaglutide Placebo
Number analyzed (Participants) | 392 | 394
Ratio of albumin | 0.99 (5.4) | 1.00 (5.2)

46. Secondary Outcome: Change in Biochemistry Parameter- Calcium
Description: Change from baseline (week 0) to week 52 in calcium (mmol/L) is presented as ratio to baseline. Results are based on the 'on-treatment' observation period which started at the date of first dose of trial product and include the period after initiation of rescue medication, if any and excludes the period after premature trial product discontinuation, if any.
Time Frame: Week 0, week 52
Population: as for outcome 32
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of calcium
Arm/Group | Semaglutide + Canagliflozin Placebo | Canagliflozin + Semaglutide Placebo
Number analyzed (Participants) | 392 | 394
Ratio of calcium | 1.01 (4.5) | 1.02 (4.1)

47. Secondary Outcome: Change in Biochemistry Parameter- Potassium
Description: Change from baseline (week 0) to week 52 in potassium (mmol/L) is presented as ratio to baseline. Results are based on the 'on-treatment' observation period which started at the date of first dose of trial product and include the period after initiation of rescue medication, if any and excludes the period after premature trial product discontinuation, if any.
Time Frame: Week 0, week 52
Population: as for outcome 32
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of potassium
Arm/Group | Semaglutide + Canagliflozin Placebo | Canagliflozin + Semaglutide Placebo
Number analyzed (Participants) | 392 | 394
Ratio of potassium | 1.00 (9.3) | 1.00 (8.6)

48. Secondary Outcome: Change in Biochemistry Parameter- Sodium
Description: Change from baseline (week 0) to week 52 in sodium (mmol/L) is presented as ratio to baseline. Results are based on the 'on-treatment' observation period which started at the date of first dose of trial product and include the period after initiation of rescue medication, if any and excludes the period after premature trial product discontinuation, if any.
Time Frame: Week 0, week 52
Population: as for outcome 32
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of sodium
Arm/Group | Semaglutide + Canagliflozin Placebo | Canagliflozin + Semaglutide Placebo
Number analyzed (Participants) | 392 | 394
Ratio of sodium | 1.00 (1.6) | 1.00 (1.5)

49. Secondary Outcome: Change in Calcitonin
Description: Change from baseline (week 0) to week 52 in calcitonin (nanograms per liter) is presented as ratio to baseline. Results are based on the 'on-treatment' observation period which started at the date of first dose of trial product and include the period after initiation of rescue medication, if any and excludes the period after premature trial product discontinuation, if any.
Time Frame: Week 0, week 52
Population: as for outcome 32
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of calcitonin
Arm/Group | Semaglutide + Canagliflozin Placebo | Canagliflozin + Semaglutide Placebo
Number analyzed (Participants) | 392 | 394
Ratio of calcitonin | 1.08 (43.8) | 1.04 (35.6)

50. Secondary Outcome: Change in Pulse
Description: Change from baseline (week 0) to week 52 in pulse is presented based on the 'on-treatment' observation period which started at the date of first dose of trial product and include the period after initiation of rescue medication, if any and excludes the period after premature trial product discontinuation, if any.
Time Frame: Week 0, week 52
Population: as for outcome 32
Measure: Mean (Standard Deviation); unit: Beats per minute (beats/min)
Arm/Group | Semaglutide + Canagliflozin Placebo | Canagliflozin + Semaglutide Placebo
Number analyzed (Participants) | 392 | 394
Beats per minute (beats/min) | 2.7 (9.5) | -0.6 (8.6)

51. Secondary Outcome: Change in ECG
Description: The electrocardiogram (ECG) was assessed by the investigator at baseline (week 0) and week 52 and categorised as normal, abnormal NCS or abnormal CS. Number of participants in each ECG category at baseline and week 52 were presented. Results are based on the 'on-treatment' observation period which started at the date of first dose of trial product and include the period after initiation of rescue medication, if any and excludes the period after premature trial product discontinuation, if any.
Time Frame: Week 0, week 52
Population: as for outcome 32
Measure: Count of Participants; unit: Participants
Arm/Group | Semaglutide + Canagliflozin Placebo | Canagliflozin + Semaglutide Placebo
Number analyzed (Participants) | 392 | 394
Participants
  Normal (week 0) | 263 | 277
  Abnormal NCS (week 0) | 126 | 117
  Abnormal CS (week 0) | 3 | 0
  Normal (week 52): number analyzed (Participants) | 331 | 340
  Normal (week 52) | 222 | 242
  Abnormal NCS (week 52): number analyzed (Participants) | 331 | 340
  Abnormal NCS (week 52) | 109 | 95
  Abnormal CS (week 52): number analyzed (Participants) | 331 | 340
  Abnormal CS (week 52) | 0 | 3

52. Secondary Outcome: Change in Physical Examination
Description: Physical examination parameters are categorised as general appearance; nervous system (central and peripheral); cardiovascular system; gastrointestinal system; skin; respiratory system; lymph node palpation; thyroid gland; left foot; right foot; left leg and right leg. The number of participants assessed as normal, abnormal not clinically significant (NCS) and abnormal clinically significant (CS) at baseline (week -2) and week 52 is presented based on the 'on-treatment' observation period which started at the date of first dose of trial product and include the period after initiation of rescue medication, if any and excludes the period after premature trial product discontinuation, if any.
Time Frame: Week -2, week 52
Population: as for outcome 32
Measure: Count of Participants; unit: Participants
Arm/Group | Semaglutide + Canagliflozin Placebo | Canagliflozin + Semaglutide Placebo
Number analyzed (Participants) | 392 | 394
Participants
  General Appearance (week -2) Normal | 345 | 335
  General Appearance (week -2) Abnormal NCS | 46 | 56
  General Appearance (week -2) Abnormal CS | 1 | 3
  General Appearance (week 52) Normal: number analyzed (Participants) | 326 | 339
  General Appearance (week 52) Normal | 294 | 304
  General Appearance (week 52) Abnormal NCS: number analyzed (Participants) | 326 | 339
  General Appearance (week 52) Abnormal NCS | 30 | 33
  General Appearance (week 52) Abnormal CS: number analyzed (Participants) | 326 | 339
  General Appearance (week 52) Abnormal CS | 2 | 2
  Nervous System (week -2) Normal: number analyzed (Participants) | 391 | 394
  Nervous System (week -2) Normal | 360 | 370
  Nervous System (week -2) Abnormal NCS: number analyzed (Participants) | 391 | 394
  Nervous System (week -2) Abnormal NCS | 26 | 21
  Nervous System (week -2) Abnormal CS: number analyzed (Participants) | 391 | 394
  Nervous System (week -2) Abnormal CS | 5 | 3
  Nervous System (week 52) Normal: number analyzed (Participants) | 326 | 339
  Nervous System (week 52) Normal | 303 | 325
  Nervous System (week 52) Abnormal NCS: number analyzed (Participants) | 326 | 339
  Nervous System (week 52) Abnormal NCS | 21 | 12
  Nervous System (week 52) Abnormal CS: number analyzed (Participants) | 326 | 339
  Nervous System (week 52) Abnormal CS | 2 | 2
  Cardiovascular System (week-2) Normal | 376 | 386
  Cardiovascular System (week -2) Abnormal NCS | 15 | 8
  Cardiovascular System (week -2) Abnormal CS | 1 | 0
  Cardiovascular System (week52) Normal: number analyzed (Participants) | 326 | 339
  Cardiovascular System (week52) Normal | 318 | 333
  Cardiovascular System (week 52) Abnormal NCS: number analyzed (Participants) | 326 | 339
  Cardiovascular System (week 52) Abnormal NCS | 7 | 6
  Cardiovascular System (week 52) Abnormal CS: number analyzed (Participants) | 326 | 339
  Cardiovascular System (week 52) Abnormal CS | 1 | 0
  Gastrointestinal System (week -2) Normal | 369 | 377
  Gastrointestinal System (week -2) Abnormal NCS | 22 | 16
  Gastrointestinal System (week -2) Abnormal CS | 1 | 1
  Gastrointestinal System (week 52) Normal: number analyzed (Participants) | 326 | 339
  Gastrointestinal System (week 52) Normal | 319 | 331
  Gastrointestinal System (week 52) Abnormal NCS: number analyzed (Participants) | 326 | 339
  Gastrointestinal System (week 52) Abnormal NCS | 7 | 8
  Gastrointestinal System (week 52) Abnormal CS: number analyzed (Participants) | 326 | 339
  Gastrointestinal System (week 52) Abnormal CS | 0 | 0
  Skin (week -2) Normal | 330 | 323
  Skin (week -2) Abnormal NCS | 62 | 69
  Skin (week -2) Abnormal CS | 0 | 2
  Skin (week 52) Normal: number analyzed (Participants) | 326 | 339
  Skin (week 52) Normal | 286 | 298
  Skin (week 52) Abnormal NCS: number analyzed (Participants) | 326 | 339
  Skin (week 52) Abnormal NCS | 39 | 40
  Skin (week 52) Abnormal CS: number analyzed (Participants) | 326 | 339
  Skin (week 52) Abnormal CS | 1 | 1
  Respiratory System (week -2) Normal | 383 | 391
  Respiratory System (week -2) Abnormal NCS | 7 | 3
  Respiratory System (week -2) Abnormal CS | 2 | 0
  Respiratory System (week 52) Normal: number analyzed (Participants) | 326 | 339
  Respiratory System (week 52) Normal | 321 | 336
  Respiratory System (week 52) Abnormal NCS: number analyzed (Participants) | 326 | 339
  Respiratory System (week 52) Abnormal NCS | 4 | 3
  Respiratory System (week 52) Abnormal CS: number analyzed (Participants) | 326 | 339
  Respiratory System (week 52) Abnormal CS | 1 | 0
  Lymph Node Palpation (week -2) Normal: number analyzed (Participants) | 391 | 394
  Lymph Node Palpation (week -2) Normal | 390 | 392
  Lymph Node Palpation (week -2) Abnormal NCS: number analyzed (Participants) | 391 | 394
  Lymph Node Palpation (week -2) Abnormal NCS | 1 | 2
  Lymph Node Palpation (week -2) Abnormal CS: number analyzed (Participants) | 391 | 394
  Lymph Node Palpation (week -2) Abnormal CS | 0 | 0
  Lymph Node Palpation (week 52) Normal: number analyzed (Participants) | 325 | 337
  Lymph Node Palpation (week 52) Normal | 325 | 337
  Lymph Node Palpation (week 52) Abnormal NCS: number analyzed (Participants) | 325 | 337
  Lymph Node Palpation (week 52) Abnormal NCS | 0 | 0
  Lymph Node Palpation (week 52) Abnormal CS: number analyzed (Participants) | 325 | 337
  Lymph Node Palpation (week 52) Abnormal CS | 0 | 0
  Thyroid Gland (week -2) Normal | 390 | 390
  Thyroid Gland (week -2) Abnormal NCS | 2 | 4
  Thyroid Gland (week -2) Abnormal CS | 0 | 0
  Thyroid Gland (week 52) Normal: number analyzed (Participants) | 326 | 338
  Thyroid Gland (week 52) Normal | 326 | 337
  Thyroid Gland (week 52) Abnormal NCS: number analyzed (Participants) | 326 | 338
  Thyroid Gland (week 52) Abnormal NCS | 0 | 1
  Thyroid Gland (week 52) Abnormal CS: number analyzed (Participants) | 326 | 338
  Thyroid Gland (week 52) Abnormal CS | 0 | 0
  Left foot (week -2) Normal | 343 | 345
  Left foot (week -2) Abnormal NCS | 47 | 44
  Left foot (week -2) Abnormal CS | 2 | 5
  Left foot (week 52) Normal: number analyzed (Participants) | 326 | 339
  Left foot (week 52) Normal | 293 | 303
  Left foot (week 52) Abnormal NCS: number analyzed (Participants) | 326 | 339
  Left foot (week 52) Abnormal NCS | 32 | 34
  Left foot (week 52) Abnormal CS: number analyzed (Participants) | 326 | 339
  Left foot (week 52) Abnormal CS | 1 | 2
  Right foot (week -2) Normal | 344 | 348
  Right foot (week -2) Abnormal NCS | 45 | 42
  Right foot (week -2) Abnormal CS | 3 | 4
  Right foot (week 52) Normal: number analyzed (Participants) | 326 | 339
  Right foot (week 52) Normal | 289 | 304
  Right foot (week 52) Abnormal NCS: number analyzed (Participants) | 326 | 339
  Right foot (week 52) Abnormal NCS | 34 | 32
  Right foot (week 52) Abnormal CS: number analyzed (Participants) | 326 | 339
  Right foot (week 52) Abnormal CS | 3 | 3
  Left leg (week -2) Normal | 348 | 358
  Left leg (week -2) Abnormal NCS | 40 | 30
  Left leg (week -2) Abnormal CS | 4 | 6
  Left leg (week 52) Normal: number analyzed (Participants) | 326 | 339
  Left leg (week 52) Normal | 300 | 314
  Left leg (week 52) Abnormal NCS: number analyzed (Participants) | 326 | 339
  Left leg (week 52) Abnormal NCS | 22 | 22
  Left leg (week 52) Abnormal CS: number analyzed (Participants) | 326 | 339
  Left leg (week 52) Abnormal CS | 4 | 3
  Right leg (week -2) Normal | 350 | 357
  Right leg (week -2) Abnormal NCS | 37 | 30
  Right leg (week -2) Abnormal CS | 5 | 7
  Right leg (week 52) Normal: number analyzed (Participants) | 326 | 339
  Right leg (week 52) Normal | 301 | 315
  Right leg (week 52) Abnormal NCS: number analyzed (Participants) | 326 | 339
  Right leg (week 52) Abnormal NCS | 19 | 21
  Right leg (week 52) Abnormal CS: number analyzed (Participants) | 326 | 339
  Right leg (week 52) Abnormal CS | 6 | 3

53. Secondary Outcome: Eye Examination
Description: Fundus photography or a dilated fundoscopy was performed by the investigator at baseline (week 0) and week 52. The results of the examination were interpreted for each eye (left/right) are categorised as normal, abnormal NCS or abnormal CS. Number of participants in each category at baseline and week 52 were presented. Results are based on the 'on-treatment' observation period which started at the date of first dose of trial product and include the period after initiation of rescue medication, if any and excludes the period after premature trial product discontinuation, if any.
Time Frame: Week 0, week 52
Population: as for outcome 32
Measure: Count of Participants; unit: Participants
Arm/Group | Semaglutide + Canagliflozin Placebo | Canagliflozin + Semaglutide Placebo
Number analyzed (Participants) | 392 | 394
Participants
  Left eye: Normal (week 0): number analyzed (Participants) | 392 | 393
  Left eye: Normal (week 0) | 322 | 319
  Left eye: Abnormal NCS (week 0): number analyzed (Participants) | 392 | 393
  Left eye: Abnormal NCS (week 0) | 65 | 71
  Left eye: Abnormal CS (week 0): number analyzed (Participants) | 392 | 393
  Left eye: Abnormal CS (week 0) | 5 | 3
  Left eye: Normal (week 52): number analyzed (Participants) | 268 | 270
  Left eye: Normal (week 52) | 231 | 228
  Left eye: Abnormal NCS (week 52): number analyzed (Participants) | 268 | 270
  Left eye: Abnormal NCS (week 52) | 30 | 40
  Left eye: Abnormal CS (week 52): number analyzed (Participants) | 268 | 270
  Left eye: Abnormal CS (week 52) | 7 | 2
  Right eye: Normal (week 0): number analyzed (Participants) | 392 | 393
  Right eye: Normal (week 0) | 321 | 319
  Right eye: Abnormal NCS (week 0): number analyzed (Participants) | 392 | 393
  Right eye: Abnormal NCS (week 0) | 66 | 70
  Right eye: Abnormal CS (week 0): number analyzed (Participants) | 392 | 393
  Right eye: Abnormal CS (week 0) | 5 | 4
  Right eye: Normal (week 52): number analyzed (Participants) | 268 | 270
  Right eye: Normal (week 52) | 225 | 226
  Right eye: Abnormal NCS (week 52): number analyzed (Participants) | 268 | 270
  Right eye: Abnormal NCS (week 52) | 35 | 44
  Right eye: Abnormal CS (week 52): number analyzed (Participants) | 268 | 270
  Right eye: Abnormal CS (week 52) | 8 | 0

54. Secondary Outcome: Total Number of Treatment-emergent Severe or Blood Glucose-confirmed Symptomatic Hypoglycaemic Episodes
Description: Hypoglycaemic episodes defined as treatment-emergent if the onset of the episode occurs within the on-treatment observation period. Severe or BG-confirmed symptomatic hypoglycaemia is an episode that is severe according to the American Diabetes Association classification or blood glucose-confirmed by a plasma glucose value <3.1 mmol/L (56 mg/dL) with symptoms consistent with hypoglycaemia. Results are based on the 'on-treatment' observation period which started at the date of first dose of trial product and include the period after initiation of rescue medication, if any and excludes the period after premature trial product discontinuation, if any.
Time Frame: Weeks 0-57
Population: Safety analysis set comprised of participants exposed to at least one dose of trial product.
Measure: Number; unit: Episodes
Arm/Group | Semaglutide + Canagliflozin Placebo | Canagliflozin + Semaglutide Placebo
Number analyzed (Participants) | 392 | 394
Episodes | 25 | 6

55. Secondary Outcome: Participants With Treatment-emergent Severe or Blood Glucose-confirmed Symptomatic Hypoglycaemic Episodes
Description: Number of participants with treatment emergent severe or blood glucose-confirmed symptomatic hypoglycaemic episodes. Hypoglycaemic episodes defined as treatment-emergent if the onset of the episode occurs within the on-treatment observation period. Severe or BG-confirmed symptomatic hypoglycaemia is an episode that is severe according to the American Diabetes Association classification or blood glucose-confirmed by a plasma glucose value <3.1 mmol/L (56 mg/dL) with symptoms consistent with hypoglycaemia. Results are based on the 'on-treatment' observation period which started at the date of first dose of trial product and include the period after initiation of rescue medication, if any and excludes the period after premature trial product discontinuation, if any.
Time Frame: Weeks 0-57
Population: Safety analysis set comprised of participants exposed to at least one dose of trial product.
Measure: Number; unit: Participants
Arm/Group | Semaglutide + Canagliflozin Placebo | Canagliflozin + Semaglutide Placebo
Number analyzed (Participants) | 392 | 394
Participants | 6 | 5

56. Secondary Outcome: Change in Short Form 36 Health Survey (SF-36): Sub-domains
Description: SF-36 is a 36-item patient-reported survey of patient health that measures the participant's overall health-related quality of life (HRQoL). SF-36v2™ questionnaire measured the HRQoL on 8 domains on individual scale ranges. The scores 0-100 (where higher scores indicated a better HRQoL) from the SF-36 were converted to norm-based scores to enable a direct interpretation in relation to the distribution of the scores in the 2009 U.S. general population. A norm-based score of 50 corresponds to the mean score and 10 corresponds to the standard deviation of the 2009 U.S. general population. Change from baseline (week 0) to week 52 in the sub-domain scores is presented. A positive change score indicate an improvement since baseline. Results are based on the 'on-treatment without rescue medication' observation period.
Time Frame: Week 0, week 52
Population: Full analysis set comprised of all randomised participants. "Number analyzed"=participants with available data.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Semaglutide + Canagliflozin Placebo | Canagliflozin + Semaglutide Placebo
Number analyzed (Participants) | 394 | 394
Score on a scale
  Physical Functioning: number analyzed (Participants) | 262 | 277
  Physical Functioning | 1.9 (7.1) | 2.7 (6.7)
  Role-physical: number analyzed (Participants) | 262 | 277
  Role-physical | 1.8 (7.3) | 2.0 (7.1)
  Bodily pain: number analyzed (Participants) | 262 | 277
  Bodily pain | 2.5 (8.9) | 1.5 (8.7)
  General health: number analyzed (Participants) | 262 | 277
  General health | 3.7 (7.7) | 3.5 (8.5)
  Social functioning: number analyzed (Participants) | 262 | 277
  Social functioning | 1.1 (8.6) | 1.1 (8.0)
  Role-emotional: number analyzed (Participants) | 262 | 277
  Role-emotional | 0.8 (9.2) | 1.2 (8.6)
  Vitality: number analyzed (Participants) | 262 | 277
  Vitality | 3.0 (8.2) | 2.0 (8.2)
  Mental health: number analyzed (Participants) | 262 | 277
  Mental health | 1.5 (8.3) | 0.6 (8.1)

57. Secondary Outcome: Change in SF-36: Physical Component Summary (PCS)
Description: Change from baseline (week 0) to week 52 in short form 36 v2.0 acute domain PCS. SF-36v2™ questionnaire measured the HRQoL on 8 domains on individual scale ranges. It consists of 2 component summary measures that further summarize 8 health domain scales. The PCS measure is derived from domain scales of physical functioning, role-physical, bodily pain, and general health. The scores 0-100 (where higher scores indicated a better HRQoL) from the SF-36 were converted to norm-based scores to enable a direct interpretation in relation to the distribution of the scores in the 2009 U.S. general population. A norm-based score of 50 corresponds to the mean score and 10 corresponds to the standard deviation of the 2009 U.S. general population. A positive change score indicates an improvement since baseline. Results are based on the 'on-treatment without rescue medication' observation period.
Time Frame: Week 0, week 52
Population: Full analysis set comprised of all randomised participants. "Number analyzed"=participants with available data.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Semaglutide + Canagliflozin Placebo | Canagliflozin + Semaglutide Placebo
Number analyzed (Participants) | 394 | 394
Score on a scale | 2.7 (6.7) | 2.9 (6.2)

58. Secondary Outcome: Change in SF-36: Mental Component Summary (MCS)
Description: Change from baseline (week 0) to week 52 in short form 36 v2.0 acute domain MCS. SF- 36v2™ questionnaire measured the HRQoL on 8 domains on individual scale ranges. The MCS measure is derived from domain scales of vitality, social functioning, role emotional and mental health. The scores 0-100 (where higher scores indicated a better HRQoL) from the SF-36 were converted to norm-based scores to enable a direct interpretation in relation to the distribution of the scores in the 2009 U.S. general population. A norm-based score of 50 corresponds to the mean score and 10 corresponds to the standard deviation of the 2009 U.S. general population. A positive change score indicates an improvement since baseline. Results are based on the 'on-treatment without rescue medication' observation period.
Time Frame: Week 0, week 52
Population: Full analysis set comprised of all randomised participants. "Number analyzed"=participants with available data.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Semaglutide + Canagliflozin Placebo | Canagliflozin + Semaglutide Placebo
Number analyzed (Participants) | 394 | 394
Score on a scale | 1.1 (8.8) | 0.5 (8.0)

59. Secondary Outcome: Change in Diabetes Treatment Satisfaction Questionnaire (DTSQ): Treatment Satisfaction Summary Score (Sum of 6 of 8 Items) and the 8 Items Separately
Description: Change from baseline (week 0) in DTSQ was evaluated at week 52. The DTSQs items are scored on a 7-point graded response scale ranging from 6 to 0. Higher scores indicate higher levels of treatment satisfaction for DTSQs items 1, 4 -8. For items 2 and 3 a higher score indicates a higher patient perceived experience of high blood sugars and low blood sugars, respectively. Thus, lower scores indicate a perception of blood glucose levels being "none of the time" unacceptably high (item 2) or low (item 3). The domain score of total treatment satisfaction (total treatment satisfaction score) was computed by adding the six items scores 1, 4-8. The score ranges 0-36. A higher treatment satisfaction score indicates a higher level of treatment satisfaction. Results are based on the 'on-treatment without rescue medication' observation period.
Time Frame: Week 0, week 52
Population: Full analysis set comprised of all randomised participants. "Number analyzed"=participants with available data.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Semaglutide + Canagliflozin Placebo | Canagliflozin + Semaglutide Placebo
Number analyzed (Participants) | 394 | 394
Score on a scale
  1) Satisfaction with treatment: number analyzed (Participants) | 263 | 280
  1) Satisfaction with treatment | 1.4 (1.6) | 1.0 (1.6)
  2) Feeling of unacceptably high blood sugars: number analyzed (Participants) | 263 | 280
  2) Feeling of unacceptably high blood sugars | -2.0 (2.2) | -1.8 (2.2)
  3) Feeling of unacceptably low blood sugars: number analyzed (Participants) | 263 | 280
  3) Feeling of unacceptably low blood sugars | 0.1 (1.9) | 0.1 (1.6)
  4) Convenience of treatment: number analyzed (Participants) | 263 | 280
  4) Convenience of treatment | 0.8 (1.8) | 0.7 (1.8)
  5) Flexibility of current treatment: number analyzed (Participants) | 263 | 280
  5) Flexibility of current treatment | 0.8 (1.7) | 0.7 (1.7)
  6) Satisfaction with understanding of diabetes: number analyzed (Participants) | 263 | 280
  6) Satisfaction with understanding of diabetes | 0.8 (1.5) | 0.6 (1.3)
  7) Recommending treatment to others: number analyzed (Participants) | 263 | 280
  7) Recommending treatment to others | 0.9 (1.5) | 0.9 (1.5)
  8) Satisfaction to continue with present treatment: number analyzed (Participants) | 263 | 280
  8) Satisfaction to continue with present treatment | 1.1 (1.8) | 0.8 (1.8)
  Total treatment satisfaction score: number analyzed (Participants) | 263 | 280
  Total treatment satisfaction score | 5.8 (7.0) | 4.8 (7.2)

60. Secondary Outcome: Change in Control of Eating Questionnaire (CoEQ): Domains
Description: The CoEQ comprised 19 items to assess the intensity and type of food cravings, as well as subjective sensation of appetite and mood, with the 4 domains: 'craving control', 'craving for sweet', 'craving for savoury' and 'positive mood'. The 19 items were scored on an 11-point graded response scale ranging from 10 to 0, with items relating to each of the 4 domains being averaged to create a final score. A low score in the domains 'craving for sweet and 'craving for savoury' represents a low level of craving; whereas a high score in the domains 'craving control' and 'positive mood' represents good control and a good mood, respectively. Results are based on the 'on-treatment without rescue medication' observation period.
Time Frame: Week 0, week 52
Population: Full analysis set comprised of all randomised participants. "Number analyzed"=participants with available data.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Semaglutide + Canagliflozin Placebo | Canagliflozin + Semaglutide Placebo
Number analyzed (Participants) | 394 | 394
Score on a scale
  Craving control: number analyzed (Participants) | 262 | 279
  Craving control | 1.0 (2.1) | 1.0 (2.5)
  Craving for sweet: number analyzed (Participants) | 262 | 279
  Craving for sweet | -0.6 (2.2) | -0.6 (2.1)
  Craving for savoury: number analyzed (Participants) | 262 | 279
  Craving for savoury | -1.1 (2.0) | -0.9 (2.0)
  Positive mood: number analyzed (Participants) | 262 | 279
  Positive mood | 0.7 (1.7) | 0.4 (1.6)

61. Secondary Outcome: Change in CoEQ: Individual Items
Description: as for outcome 60
Time Frame: Week 0, week 52
Population: Full analysis set comprised of all randomised participants. "Number analyzed"=participants with available data.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Semaglutide + Canagliflozin Placebo | Canagliflozin + Semaglutide Placebo
Number analyzed (Participants) | 394 | 394
Score on a scale
  How hungry have you felt: number analyzed (Participants) | 262 | 279
  How hungry have you felt | -1.2 (2.6) | -0.8 (2.6)
  How full have you felt: number analyzed (Participants) | 262 | 279
  How full have you felt | 0.2 (2.7) | 0.0 (2.7)
  How often have you had cravings (last 7 days): number analyzed (Participants) | 262 | 279
  How often have you had cravings (last 7 days) | -0.9 (2.9) | -1.1 (3.0)
  How strong have any cravings been: number analyzed (Participants) | 262 | 279
  How strong have any cravings been | -0.9 (2.9) | -1.1 (3.0)
  Difficulty to resist cravings: number analyzed (Participants) | 262 | 279
  Difficulty to resist cravings | -0.9 (2.9) | -0.8 (3.2)
  Ate in response to cravings: number analyzed (Participants) | 262 | 279
  Ate in response to cravings | -0.9 (2.7) | -0.7 (3.2)
  Difficulty to control eating: number analyzed (Participants) | 262 | 279
  Difficulty to control eating | -1.5 (2.8) | -1.2 (3.0)
  Desire to eat savory food: number analyzed (Participants) | 262 | 279
  Desire to eat savory food | -1.4 (2.6) | -1.0 (2.8)
  Craving for dairy foods: number analyzed (Participants) | 262 | 279
  Craving for dairy foods | -0.8 (2.9) | -0.6 (3.1)
  Craving for starchy foods: number analyzed (Participants) | 262 | 279
  Craving for starchy foods | -1.4 (2.7) | -1.1 (3.0)
  Craving for savory foods: number analyzed (Participants) | 262 | 279
  Craving for savory foods | -0.9 (2.9) | -0.9 (2.9)
  Desire to eat sweet food: number analyzed (Participants) | 262 | 279
  Desire to eat sweet food | -0.9 (3.1) | -1.0 (2.9)
  Craving for chocolate: number analyzed (Participants) | 262 | 279
  Craving for chocolate | -0.3 (3.1) | -0.4 (2.9)
  Craving for other sweets: number analyzed (Participants) | 262 | 279
  Craving for other sweets | -0.6 (2.8) | -0.6 (2.8)
  Craving for fruit or fruit juice: number analyzed (Participants) | 262 | 279
  Craving for fruit or fruit juice | -0.6 (3.0) | -0.6 (3.2)
  Felt happy: number analyzed (Participants) | 262 | 279
  Felt happy | 0.8 (2.5) | 0.4 (2.3)
  Felt anxious: number analyzed (Participants) | 262 | 279
  Felt anxious | -0.9 (3.1) | -0.6 (2.7)
  Felt alert: number analyzed (Participants) | 262 | 279
  Felt alert | 0.2 (2.4) | 0.0 (2.4)
  Felt contented: number analyzed (Participants) | 262 | 279
  Felt contented | 0.8 (2.4) | 0.5 (2.2)

ADVERSE EVENTS:
Time Frame: From the date of first dose of trial product (week 0) to end of treatment (week 52) + post treatment follow-up of 5 weeks.
Description: Evaluation of safety was based on SAS which comprised of all randomised participants who received at least one dose of trial product.
  AEs with onset during the on-treatment observation period (the period when participants were exposed to trial product) were considered treatment-emergent.
Arm/Group | Semaglutide + Canagliflozin Placebo | Canagliflozin + Semaglutide Placebo
All-Cause Mortality (participants affected / at risk) | 1/392 | 0/394
Serious Adverse Events (participants affected / at risk) | 18/392 | 21/394
Other Adverse Events (participants affected / at risk) | 185/392 | 120/394
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Semaglutide + Canagliflozin Placebo (N=392) | Canagliflozin + Semaglutide Placebo (N=394)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0)
Airway complication of anaesthesia (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Angina unstable (Cardiac disorders) | 0 (0) | 1 (1)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Aphasia (Nervous system disorders) | 1 (1) | 0 (0)
Arteriosclerosis (Vascular disorders) | 1 (1) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 1 (1)
Bartholin's cyst (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Basal ganglia haemorrhage (Nervous system disorders) | 0 (0) | 1 (1)
Bipolar disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Cataract (Eye disorders) | 1 (1) | 0 (0)
Cellulitis gangrenous (Infections and infestations) | 0 (0) | 1 (1)
Cellulitis staphylococcal (Infections and infestations) | 0 (0) | 1 (1)
Chest pain (General disorders) | 0 (0) | 1 (1)
Cholecystitis chronic (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 3 (3)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Confusional state (Psychiatric disorders) | 1 (1) | 0 (0)
Coronary artery disease (Cardiac disorders) | 0 (0) | 1 (1)
Coronary artery stenosis (Cardiac disorders) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Glomerular filtration rate decreased (Investigations) | 1 (1) | 0 (0)
Haemorrhoids thrombosed (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hepatic cirrhosis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hydronephrosis (Renal and urinary disorders) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 1 (1) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Myocardial ischaemia (Cardiac disorders) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 2 (2) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (2) | 1 (1)
Patella fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Perirectal abscess (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 1 (1)
Post procedural haematuria (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Prescribed overdose (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Prostatism (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 2 (2)
Respiratory tract infection viral (Infections and infestations) | 0 (0) | 1 (1)
Retinal infarction (Eye disorders) | 1 (1) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Splenomegaly (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Transaminases increased (Investigations) | 0 (0) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 1 (1)
Ureterolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 3 (3) | 0 (0)
Urosepsis (Infections and infestations) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Vulval abscess (Infections and infestations) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Semaglutide + Canagliflozin Placebo (N=392) | Canagliflozin + Semaglutide Placebo (N=394)
Back pain (Musculoskeletal and connective tissue disorders) | 11 (11) | 21 (21)
Constipation (Gastrointestinal disorders) | 20 (20) | 23 (23)
Decreased appetite (Metabolism and nutrition disorders) | 26 (26) | 6 (6)
Diarrhoea (Gastrointestinal disorders) | 59 (94) | 37 (58)
Dyspepsia (Gastrointestinal disorders) | 22 (23) | 8 (8)
Headache (Nervous system disorders) | 26 (48) | 27 (47)
Nasopharyngitis (Infections and infestations) | 23 (25) | 26 (34)
Nausea (Gastrointestinal disorders) | 89 (127) | 26 (30)
Vomiting (Gastrointestinal disorders) | 50 (77) | 9 (9)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
At the end of the trial, one or more scientific publications may be prepared collaboratively by the investigator(s) and Novo Nordisk. Novo Nordisk reserves the right to postpone publication and/or communication for up to 60 days to protect intellectual property.

DOCUMENTS (2):
  • Study Protocol (2019-06-03): https://cdn.clinicaltrials.gov/large-docs/84/NCT03136484/Prot_000.pdf
  • Statistical Analysis Plan (2019-06-03): https://cdn.clinicaltrials.gov/large-docs/84/NCT03136484/SAP_001.pdf